CLINICAL TRIAL: NCT02819154
Title: Study of the Social and Psychological Consequences of ICU Hospitalization
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: SEPPICC
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2016-06

CONDITIONS: Intensive Care Units

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: phone call to evaluate the social changes, emotional, professional a cohort of patients following ICU stay — phone call to evaluate the social changes, emotional, professional a cohort of patients following ICU stay. Investigators will use :
  * Questionnaire SF 36: Only the first two questions of the SF-36 are used exploring the felt quality of life at the time of the telephone call and in comparison with the period before hospitalization in intensive care.
  * Stress Assessment Questionnaire posttraumatic (Revised Impact of Event Scale, IES-R)
  * ADL: Assessment of independence in activities of daily life

SUMMARY:
Patients are admitted to intensive care for serious diseases (sepsis, ARDS ...) burdened with a high mortality rate. Invasive methods of resuscitation and the diseases treated can lead to serious sequelae. Follow-up studies of patients at hospital discharge report most often the quality of life using validated quantitative scales. A recent consensus of the American Society of resuscitation an update on the physical, cognitive and psychological sequelae of ICU hospitalization for the family and the patient, grouped under the term "post-intensive care syndrome." Social changes, emotional and professional are little studied and are not part of the information provided by the quality of life questionnaires. The investigators hypothesize that intensive care stay entails a profound effect on the lives of patients. This study will add additional data on a little known aspect of post resuscitation.

DETAILED DESCRIPTION:
Primary objective :

To evaluate the social changes, emotional, professional a cohort of patients following ICU stay

Secondary objective:

Evaluate post traumatic stress disorder and quality of life of a cohort of patients following ICU stay

Methods :

Study design Study of bi-center cohort (ICUs of Saint Joseph and Bichat hospitals).

prospective follow the consequences of the intensive use of patient already included in the Outcomerea database using quality of life questionnaires, independence and post-traumatic stress and a questionnaire constructed for the study.

Patient selection in the database The database contains more than 10,000 visits. Investigators will select the patients in the two hospitals in the study. Then a second selection will be based on the inclusion criteria. The review of hospital records will not include patients with the first five criteria for non-inclusion. These patients appear in the flow chart

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted in ICU and who had at least one organ dysfunction (need at least 24 hours of mechanical ventilation) in two intensive care units

Exclusion Criteria:

* Patient Do not speak French
* Patient aphasic deaf
* Patient with xxistencing cognitive disorders
* Homeless

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient admitted in ICU and who had at least one organ dysfunction (need at least 24 hours of mechanical ventilation) in two intensive care units
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-10-24 (Actual); Primary Completion 2016-05-30 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Assessment of change of Life quality with SP 36 questionnary | Day 0 at the end of hospitalization, 6 months after hospitalization
  Only the first two questions of the SF-36 are used exploring the felt quality of life at the time of the telephone call and in comparison with the period before hospitalization in intensive care.

SECONDARY OUTCOMES:
Stress Assessment Questionnaire posttraumatic | Day 0 at the end of hospitalization, 6 months after hospitalization
  Stress Assessment Questionnaire posttraumatic (Revised Impact of Event Scale, IES-R)
Assessment of independence in activities of daily life | Day 0 at the end of hospitalization, 6 months after hospitalization
  ADL: Assessment of independence in activities of daily life

CONTACTS AND LOCATIONS:
Overall Officials: GARROUSTE Maite, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France